CLINICAL TRIAL: NCT04754464
Title: Randomised, Controlled, Double-blind Clinical Study on the Effect of a Synbiotic on Body Fat Mass, Weight Management, Metabolic Syndrome and Other Risk Factors for CVD and Diabetes, on Fecal Microbiota and Adverse Effects
Brief Title: Clinical Study on the Effect of a Synbiotic on Body Fat Mass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Slimbiotics GmbH (Industry)
Collaborators: Clinical Research Center Kiel GmbH (Other)
Responsible Party: Sponsor
Organization: Slimbiotics (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Slim-LfX- 2020
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Type 2 Diabetes; Metabolic Syndrome; Obesity, Abdominal; Obesity, Visceral
Keywords: synbiotic; body fat mass; metabolic syndrome; diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome; Obesity, Abdominal; Diabetes Mellitus | interventions — Synbiotics; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: Randomised, controlled, double-blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo products are identical with verum in smell, flavour, color, texture, appearance, packaging (sachets) and labelling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- synbiotic (Active Comparator): synbiotic consisting of three different strains of Lactobacillus fermentum + acacia gum (gum arabic)
  Interventions: Dietary Supplement: synbiotic
- microcrystalline cellulose (Placebo Comparator): microcrystalline cellulose
  Interventions: Dietary Supplement: microcrystalline cellulose

INTERVENTIONS:
Dietary Supplement: synbiotic — Consumption of 6 g powder consisting of the strains Lactobacillus fermentum K7-Lb1, L. fermentum K8-Lb1, L. fermentum K11-Lb3, acacia gum (gum arabic), maltodextrin, sucralose and flavour twice a day resolved in water
  Arms: synbiotic
Dietary Supplement: microcrystalline cellulose — Consumption of 6 g powder containing microcrystalline cellulose, maltodextrin , sucralose and flavour twice a day, resolved in water
  Arms: microcrystalline cellulose

SUMMARY:
In this trial the effect of a synbiotic consisting of the three different strains of Lactobacillus fermentum and acacia gum (gum arabic) on body fat mass, body weight, long-term glycemia, insulin resistance and other risk factors for CVD and diabetes in overweight type 2 diabetics is investigated.

DETAILED DESCRIPTION:
The effects of probiotics on glucose and lipid metabolism, on body fat, weight, visceral fat and liver steatosis were shown by several meta-analyses for the total variety, as described above. Some probiotic species/strains, however, seem to be more efficacious. The lactobacilli used in this trial were selected for their anti-inflammatory properties and based on induction of defensins in enterocytes. Therefore, one may expect more pronounced effects of these strains on traits of the metabolic syndrome, which is driven by low grade inflammation, than those found in the meta-analyses for the whole variety of probiotics without discriminating species and strain specificity.

The combination of these Lactobacillus strains with acacia gum is expected to enable even more pronounce effects, since acacia gum was shown to increase the number of lactobacilli in the gut and, hence, are supposed to promote their propagation and, hence their effects. The dosage of 10 g/day acacia gum was demonstrated to be sufficient for enhancing fecal lactobacilli and bifidobacterial.

ELIGIBILITY:
Inclusion Criteria:

1. Overweight or obese (BMI ≥ 25)
2. Type 2 diabetes
3. Age ≥ 18
4. Written informed consent

Exclusion Criteria:

Any of the following is regarded as a criterion for exclusion from enrollment into the study:

1. Subjects currently enrolled in another clinical study
2. Subjects having finished another clinical study within the last 4 weeks before inclusion
3. Hypersensitivity, allergy or intolerance against any compound of the test products (e. g. acacia gum)
4. Condition after implantation of a cardiac pacemaker or other active implants
5. Antidiabetic drugs except metformin
6. Any disease or condition which might compromise significantly the hepatic (ascites), hematopoietic, renal, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal or any other body system with the exception of the conditions defined by the inclusion criteria
7. History of hepatitis B, C, HIV
8. History of or present liver deficiency as defined by Quick < 70%
9. Regular medical treatment including OTC, which may have impact on the study aims (e.g. probiotics containing supplements etc.)
10. Major cognitive or psychiatric disorders
11. Subjects who are scheduled to undergo any diagnostic intervention or hospitalization which may cause protocol deviations
12. Simultaneous study participation by members of the same household
13. Pregnancy and lactation
14. Any diet to lose body weight
15. Eating disorders or vegan diet
16. Anorexic drugs and laxatives
17. Present drug abuse or alcoholism
18. Legal incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
BFM | 12 weeks
  Body Fat Mass (BFM) as assessed by bioelectrical impedance analysis (BIA) (alteration V3-V1; verum versus placebo group)

SECONDARY OUTCOMES:
HbA1c | 12 weeks
  Glycated Hemoglobin
HOMA-IR | 12 weeks
  HOMA-IR (Homeostasis Model Assessment (HOMA)-IR = glucose [mmol/L] x insulin [µU/ml]/22,5) as parameter for insulin resistance

OTHER OUTCOMES:
WC | 12 weeks
  Waist Circumference
WHtR | 12 weeks
  waist-to-height ratio

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Laue, Dr. med., Principal Investigator — Clinical Research Center Kiel
Locations (2):
- Slimbiotics GmbH, Vienna, Austria
- Clinical Research Center Kiel, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No